CLINICAL TRIAL: NCT06572852
Title: Next-Generation Endometriosis Diagnostics Through Comprehensive Multi-Dimensional Analysis
Acronym: AdEnd
Status: Recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Collaborators: AUO Renato Dulbecco (Unknown)
Responsible Party: Principal Investigator, Candiani Massimo, Principal Investigator, IRCCS San Raffaele
Other Study IDs: PNRR-MCNT2-2023-12378346
Record Dates: First submitted 2024-08-23; First posted 2024-08-27 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-10

CONDITIONS: Endometriosis; Adenomyosis
Keywords: Case-control; Retrospective; Prospective; Genetic; Endometriosis; Adenomyosis; Machine learning; Epigenetic
MeSH Terms: conditions — Endometriosis; Adenomyosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Biospecimen Retention: Samples With DNA — The biological samples collected for the study include blood and uterine fluid.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (5):
- Cases with both endometriosis and adenomyosis: 100 women diagnosed with both endometriosis and adenomyosis (cases). These participants are part of couples seeking fertility treatment at Assisted Reproduction Centers. The diagnosis of both endometriosis and adenomyosis will be made through ultrasound imaging at the IVF centers. The recruitment involves the collection of blood for genetic and epigenetic analysis, and acquiring ultrasound images for machine learning analysis.
  Interventions: Other: No intervention
- Cases with only endometriosis: 15 women diagnosed exclusively with endometriosis (cases): This subgroup consists of women who have been diagnosed with endometriosis but show no ultrasound evidence of adenomyosis. The recruitment involves the collection of blood for genetic and epigenetic analysis, acquiring ultrasound images for machine learning analysis, and collecting uterine fluid samples to study gene expression profiles through uterine fluid extracellular vesicles (UF-EVs).
  Interventions: Other: No intervention
- Cases with only adenomyosis: 15 women diagnosed exclusively with adenomyosis (cases): This subgroup includes women diagnosed solely with adenomyosis, without any ultrasonographic signs of endometriosis. The recruitment involves the collection of blood for genetic and epigenetic analysis, acquiring ultrasound images for machine learning analysis, and collecting uterine fluid samples to study gene expression profiles through uterine fluid extracellular vesicles (UF-EVs).
  Interventions: Other: No intervention
- Controls: 400 women from couples seeking fertility treatment at infertility clinics (controls): These participants, who will be part of couples attempting to conceive, will be actively seeking treatment for infertility or other gynecological symptoms. Crucially, these individuals will have undergone ultrasound screenings that have excluded the presence of endometriosis or adenomyosis. The recruitment involves the collection of blood for genetic and epigenetic analysis, and acquiring ultrasound images for machine learning analysis.
  Interventions: Other: No intervention
- Cases of endometriosis with pre-existing genotyping data: This group will consist of 300 DNA biobanked samples from women diagnosed with endometriosis. These samples come with pre-existing genotyping data, which will be integrated into the study to provide a robust genetic baseline for comparative analyses.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
This study is a multicentric, observational, case-control, non-profit with additional procedures. It aims to deepen the understanding of the chronic gynecological conditions of endometriosis and adenomyosis, which significantly impact women's reproductive health. Its purpose is to improve early diagnosis and personalized treatment of these conditions using a multi-omic approach, that integrates genetic, epigenetic, imaging, and endometrial receptivity data. The goal is also to refine image-based predictions through recent advancements in artificial intelligence and to study uterine extracellular vesicles to assess fertility non-invasively.

The study targets patients with endometriosis and/or adenomyosis and involves women seeking fertility treatments at assisted reproduction centers, who will serve as a control population.

The study comprises both prospective and retrospective components. The prospective recruitment involves the collection of blood and uterine fluid samples, while the retrospective element utilizes pre-existing biobank samples for comprehensive genetic and epigenetic analysis.

DETAILED DESCRIPTION:
Recent research indicates that epigenetic blood analysis could revolutionize the diagnosis of endometriosis, moreover, strong correlations between endometrial and blood methylation have been reported, suggesting significant diagnostic potential. Preliminary data on Polygenic Risk Scores (PRS) also show promise in identifying genetic profiles associated with disease severity.

Advancements in artificial intelligence (AI) offer precise image-based diagnostic predictions, highlighting the transformative potential of integrating AI with genetic analyses. Additionally, our preliminary studies have demonstrated the potential of using gene expression data from uterine fluid extracellular vesicles (UF-EVs) to understand endometrial receptivity, with implications for detecting both endometriosis and adenomyosis.

Through this study, the investigators hypothesize that differential methylation profiles, integrated with genetic, epigenetic, and clinical data, can accurately classify endometriosis and adenomyosis cases. Additionally, it's hypothesized that UF-EVs gene expression profiles differ significantly between endometriosis, adenomyosis, and fertile controls, providing critical insights into endometrial receptivity and potential diagnostic markers for these conditions.

Primary Objective:

To identify specific CpG sites that exhibit differential methylation levels between endometriosis cases and controls. These methylation profiles, combined with polygenic risk scores (PRS) and clinical questionnaire data, will be used to classify cases and controls through machine learning analysis. (Aim 1) In addition to the differential methylation analysis, 'high-resolution SNP genotyping' will be employed. This genotyping will adjust the methylation analysis and aid in deriving polygenic risk scores.

Secondary Objectives:

To develop and validate a diagnostic model integrating ultrasound imaging with genetic, epigenetic, and clinical data to accurately identify and differentiate adenomyosis as an extension of endometriosis, and to predict pregnancy outcomes in women undergoing IVF. (Aim 2)

Tertiary Objectives:

To characterize the gene expression profiles of uterine fluid extracellular vesicles (UF-EVs) specific to endometriosis and adenomyosis will be analyzed samples at two critical time points: LH+2 (non-receptive) and LH+7 (receptive). The obtained gene expression data will be compared against previously collected data from fertile and infertile patients. By comparing these profiles, the investigators aim to identify distinct molecular signatures associated with each condition, enhancing our understanding of their impact on fertility and endometrial receptivity. Also, this comparison will allow us to refine diagnostic markers and potentially develop targeted interventions for affected women. (Aim 3)

This study is conducted as a multicenter project, involving two Assisted Reproduction Centers, it will include a diverse cohort of 800 women. The study involves 530 participants and three distinct groups: women diagnosed with endometriosis, women diagnosed with both endometriosis and adenomyosis, and a control group of infertile women without these conditions. Each group will participate in the study, it is planned to last 24 months from the onset of recruitment to the final analysis of collected data. An additional group will consist of 300 DNA biobanked samples from women diagnosed with endometriosis.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for cases with endometriosis and adenomyosis, must meet the following criteria:

* Able to give informed consent for participation in the study.
* European descent.
* Confirmed diagnosis of both endometriosis and adenomyosis through ultrasound screening.
* Listed for assisted reproductive treatment, specifically within their first or second IVF cycle.

Participants eligible for cases with only endometriosis must meet the following criteria:

* Able to give informed consent for participation in the study.
* European descent.
* Confirmed diagnosis of endometriosis with no ultrasound evidence of adenomyosis.
* Enrolled in an assisted reproductive treatment cycle involving embryo thawing.

Participants eligible for cases with only adenomyosis must meet the following criteria:

* Able to give informed consent for participation in the study.
* European descent.
* Confirmed diagnosis of adenomyosis with no ultrasound evidence of endometriosis.
* Enrolled in an assisted reproductive treatment cycle involving embryo thawing.

Participants eligible as controls must meet the following criteria:

* Able to give informed consent for participation in the study.
* European descent.
* Undergone ultrasound screenings that have excluded the presence of endometriosis or adenomyosis.
* Listed for assisted reproductive treatment, specifically within their first or second IVF cycle.
* Presence of reduced ovarian reserve or non-severe male factor infertility.

Exclusion Criteria:

* Patients unable or unwilling to sign the informed consent
* Individuals who exhibit the presence of sactosalpinx or other uterine pathologies such as fibroids, polyps, or irregular endometrial thickening will be excluded from participation in this study.

These exclusion criteria are applicable across all groups to ensure the accuracy and reliability of the study's findings related to endometriosis and adenomyosis.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will involve a total of 530 participants selected from two Assisted Reproduction Centers. The participant population includes:
  * Group A: 100 women diagnosed with both endometriosis and adenomyosis (cases).
  * Group B: 15 women diagnosed exclusively with endometriosis (cases).
  * Group C: 15 women diagnosed exclusively with adenomyosis (cases).
  * 400 women from couples seeking fertility treatment at infertility clinics (controls).
  Additionally, Group D will consist of 300 DNA biobank samples from women diagnosed with endometriosis.
Sampling Method: Non-Probability Sample
Enrollment: 530 (Estimated)
Dates: Start 2024-11-07 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-30 (Estimated)

PRIMARY OUTCOMES:
Identification of epigenetic profile | 2 years
  To identify specific CpG sites that exhibit differential methylation levels between endometriosis cases and controls. These methylation profiles, polygenic risk scores (PRS), and clinical questionnaire data will be used to classify cases and controls through machine learning analysis.
Identification of genetic profile | 2 years
  In addition to the differential methylation analysis, 'high-resolution SNP genotyping' will be employed. This genotyping will adjust the methylation analysis and aid in deriving polygenic risk scores.

SECONDARY OUTCOMES:
Development and validation of a diagnostic model | 2 years
  To develop and validate a diagnostic model integrating ultrasound imaging with genetic, epigenetic, and clinical data to accurately identify and differentiate adenomyosis as an extension of endometriosis, and to predict pregnancy outcomes in women undergoing IVF.

OTHER OUTCOMES:
Characterization of uterine fluid extracellular vesicles (UF-EVs) | 2 years
  To characterize the gene expression profiles of uterine fluid extracellular vesicles (UF-EVs) specific to endometriosis and adenomyosis, we will analyze samples at two critical time points: LH+2 (non-receptive) and LH+7 (receptive). We will compare the obtained gene expression data against previously collected data from fertile and infertile patients. By comparing these profiles, we aim to identify distinct molecular signatures associated with each condition, enhancing our understanding of their impact on fertility and endometrial receptivity. Also, this comparison will allow us to refine diagnostic markers and potentially develop targeted interventions for affected women.

CONTACTS AND LOCATIONS:
Overall Officials: MASSIMO CANDIANI, Principal Investigator — IRCCS San Raffaele
Locations (2):
- Italy (2):
  - Azienda Ospedaliero Universitaria Renato Dulbecco di Catanzaro, Catanzaro, Catanzaro
  - IRCCS San Raffaele Hospital, Milan, Milano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Giacomini E, Scotti GM, Vanni VS, Lazarevic D, Makieva S, Privitera L, Signorelli S, Cantone L, Bollati V, Murdica V, Tonon G, Papaleo E, Candiani M, Vigano P. Global transcriptomic changes occur in uterine fluid-derived extracellular vesicles during the endometrial window for embryo implantation. Hum Reprod. 2021 Jul 19;36(8):2249-2274. doi: 10.1093/humrep/deab123. PMID 34190319
- [Background] Vercellini P, Vigano P, Bandini V, Buggio L, Berlanda N, Somigliana E. Association of endometriosis and adenomyosis with pregnancy and infertility. Fertil Steril. 2023 May;119(5):727-740. doi: 10.1016/j.fertnstert.2023.03.018. Epub 2023 Mar 21. PMID 36948440